CLINICAL TRIAL: NCT01122121
Title: Comparative Efficacy and Safety of Combined Radiotherapy and Adjuvant Hormone Therapy (Leuprorelin SR 11.25 mg) and Hormone Therapy Alone (Leuprorelin SR 11.25 mg) in Locally Advanced Prostate Cancer (T3-T4 or pT3 on Biopsy, N0, M0)
Brief Title: Leuprorelin Associated With Radiotherapy Versus Leuprorelin Alone in T3 - T4 or pT3 (on Biopsy) N0, M0 Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP III/98/032; U1111-1169-6728 (Registry Identifier: WHO)
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Prostatic Neoplasms, Locally Advanced
Keywords: Drug Therapy; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Flutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined Radiotherapy and Hormone Therapy (Experimental): Leuprorelin 11.25 milligram (mg) sustained release (SR), injection, subcutaneously, once every 3 months up to 3 years and flutamide 250 mg, tablet, orally, thrice daily for 30 days from the first dose of leuprorelin. Radiotherapy 70 +/- 4 Gray (Gy) in 35 fractions at a rate of 5 fractions of 2 Gy per week up to 3 years. An interval of a maximum of 2 weeks is authorized between radiation of the pelvis with 50 Gy (±4) (5 weeks) and radiation of the prostate with an additional 20 Gy.
  Interventions: Drug: Leuprorelin SR; Radiation: Radiotherapy; Drug: Flutamide
- Hormone Therapy alone (Active Comparator): Leuprorelin 11.25 mg SR, injection, subcutaneously, once every 3 months up to 3 years and flutamide 250 mg, tablet, orally, thrice daily for 30 days from the first dose of leuprorelin.
  Interventions: Drug: Leuprorelin SR; Drug: Flutamide

INTERVENTIONS:
Drug: Leuprorelin SR — Leuprorelin SR injection
  Other Names: ENANTONE SR
Radiation: Radiotherapy — Radiotherapy 70 +/- 4 Gy
  Arms: Combined Radiotherapy and Hormone Therapy
Drug: Flutamide — Flutamide tablets

SUMMARY:
The purpose of this study is to compare the efficacy and safety of combined radiotherapy and hormone therapy and hormone therapy alone in the treatment of clinically locally advanced prostate cancer (T3-T4 or pT3 on biopsy, N0, M0).

DETAILED DESCRIPTION:
The drug being tested in this study is called leuprorelin SR. Leuprorelin SR is being tested to treat people who have prostate cancer. This study will look at the overall survival of people who take leuprorelin SR in addition to radiation therapy compared to those who take only leuprorelin SR.

The study will enroll approximately 273 patients. Participants will be randomly assigned to one of the two treatment groups.

* Combined Radiotherapy and Hormone Therapy
* Hormone Therapy alone. All participants will receive leuprorelin injection every 3 months and flutamide tablets thrice daily for first 30 days as part of hormone therapy. Participants randomized to combined radiotherapy and hormone therapy group, will also receive radiotherapy 70 +/- 4 Gy in 35 fractions at a rate of 5 fractions of 2 Gy per week.

This multi-center trial will be conducted in France and Tunisia. The overall time to participate in this study is 8 years. The scheduled duration of hormone therapy was 3 years in both arms, with an additional treatment-free follow-up period of 2 years i.e. a total follow-up period of 5 years. Post-protocol collection of information relative to survival will be performed after the end the 5-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced adenocarcinoma of the prostate, graded: T3 or T4 or pT3 on biopsies (presence of tumour tissue in periprostatic fat observed on biopsies), N0 (absence of metastatic), M0 (no distant metastases detectable on the following examinations: bone scan, chest x-ray, abdominal and pelvic ultrasound).
* Patient in whom the prostatic adenocarcinoma has received no prior treatment of any type, with the possible exception of transurethral resection due to obstructive symptoms.
* Patient with a Karnofsky index greater than or equal to (≥) 70.
* Patient aged under 80 years on the randomization date.
* Patient with a life expectancy of at least 7 years.
* Patient who, after having received clear information, gave his written consent to participate and cooperate in the study.
* Patient for whom a recent blood test (less than [<] 2 months) has not revealed elevated transaminases ≥ 3 times the normal laboratory range.

Exclusion Criteria:

* Patient incapable of understanding the information supplied concerning the study or of giving his consent, or having refused to sign the informed consent form,
* Patient for whom there is a risk that follow-up in compliance with the conditions stipulated by the protocol will not be possible,
* Patient having already received prior treatment for prostate cancer, excluding transurethral resection of the prostate to relieve obstruction,
* Patient having undergone surgical castration, or with a history of bilateral adrenalectomy or hypophysectomy,
* Patient having had another cancer within the previous 5 years (including carcinoma in situ of the bladder) excluding basocellular epithelioma or carcinoma in situ (other than in the bladder),
* Patient with lymph node or metastatic spread of the prostatic adenocarcinoma suspected on imaging,
* Patient with a non-controlled severe active disease,
* Patient with a contraindication to external prostatic radiotherapy,
* Patient receiving or having received another experimental treatment within 3 months prior to inclusion in the study,
* Patient with impaired liver function or elevated transaminases ≥3 times the normal laboratory range.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2000-03; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 5 years | Year 5
  PFS=time from randomization to first documentation of progression (death, biological progression or clinical progression). PFS at Year 5=probability of participants' PFS at Year 5. Biological progression definition I: halfway point between nadir and first rise with prostate-specific antigen (PSA) ≥1 nanogram per milliliter (ng/mL) signifying progression and date of introduction of prostate treatment for all participants, including those leaving prematurely for reason other than progression/death; definition II: first date when PSA=nadir+2 ng/mL and date of introduction of prostate treatment, for participants leaving prematurely for reason other than progression/death. Clinical progression: local clinical progression->50% increase in prostate volume relative to lowest volume, recurrence of palpable prostatic tumor after complete regression, positive biopsy; locoregional progression=pelvic regional lymph node lesion development; metastatic progression=distant lesions identification.

SECONDARY OUTCOMES:
Time to Biological Progression | Baseline up to Year 5
  Biological progression as per definition I is defined as halfway point between nadir and first rise with PSA greater than or equal to (≥) 1 ng/mL signifying progression and date of introduction of prostate treatment for all participants, including those leaving prematurely for reason other than progression/death; and as per definition II, it is defined as first date when PSA=nadir+2 ng/mL and date of introduction of prostate treatment, for participants leaving prematurely for reason other than progression/death. Time to onset of biological progression will be performed using the Kaplan- Meier method taking into account the date of onset of the first biological progression. The participants will be censored on the date of death, lost to follow-up or living without biological progression on the date of the last news.
Time to Clinical Progression | Baseline up to Year 5
  Clinical progression is based on three parameters: local clinical progression which is defined as greater than (>) 50 percent (%) increase in prostate volume relative to lowest volume, recurrence of palpable prostatic tumor after complete regression, positive biopsy; locoregional progression which is defined as pelvic regional lymph node lesion development; and metastatic progression which is defined as distant lesions identification. Time to onset of clinical progression will be performed using the Kaplan-Meier method based on the date of onset of the first progression among local, locoregional or metastatic clinical progressions.
Overall Survival | Baseline up to Year 5
  Overall survival will be measured as the time from the date of randomization to the date of death. Participants will be censored in case of lost to follow-up or alive on the date of the last news.
Time to Locoregional Progression | Baseline up to Year 5
  Locoregional progression is defined as the development of pelvic regional lymph node lesion(s) identified by computed tomography (CT) scan or ultrasound and confirmed by biopsy in the absence of any other signs of progression. It will be performed using the Kaplan-Meier method taking into account the date of onset of locoregional progression.
Time to Onset of Metastatic Progression | Baseline up to Year 5
  Metastatic progression is defined as identification of distant lesions. Time to onset of metastatic progression will be performed using the Kaplan-Meier method taking into account the date of onset of the first metastatic progression. The participants will be censored in case of death, lost to follow-up or alive without metastatic progression on the date of the last news.
Specific Survival | Baseline up to Year 5
  Analysis of specific survival using the Kaplan-Meier method takes into account the dates of death linked to the disease. The participants will be censored in case of death, lost to follow-up or alive on the date of the last news.
Number of Deaths linked to the disease | Baseline up to Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, Dr, Principal Investigator — Clinique Mutualiste - Saint-Etienne; Pierre RICHAUD, Dr, Principal Investigator — Institut BERGONIÉ, Centre Régional de Lutte contre le Cancer, Bordeaux; Michel PENEAU, Dr, Principal Investigator — Martinique; Jean-Jacques MAZERON, Pr, Principal Investigator — Groupe Hospitalier PITIE-SALPETRIERE, Paris
Locations (1):
- Clinique Mutualiste, Saint-Etienne, France

REFERENCES:
- [Derived] Sargos P, Mottet N, Bellera C, Richaud P. Long-term androgen deprivation, with or without radiotherapy, in locally advanced prostate cancer: updated results from a phase III randomised trial. BJU Int. 2020 Jun;125(6):810-816. doi: 10.1111/bju.14768. Epub 2020 Mar 2. PMID 30946523